CLINICAL TRIAL: NCT06351397
Title: Immersive Mixed Reality Simulation to Evoke Empathy
Acronym: Empathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 75021
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Educational Problems
Keywords: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed Reality Group (Experimental): In the MR group, the simulation instructor will explain the scope of the simulation embodiment experience and equip a weighted vest on the participant as they are asked to lay on a hospital patient gurney, seated upright. The participant, who is wearing a weighted vest to simulate an anterior mediastinal mass, will be asked to be seated upright and will view various holograms including vitals monitors, hear hospital related sounds via the headset, and also see additional holographic assets including intravenous polls and a defibrillator as well as experience heat (simulating a fever) from heat lamps. The simulation instructor will play the role of a physician who is using good communication skills based on the Calgary-Cambridge Guide to review a scripted consent for a high risk biopsy under sedation that may require life saving interventions such as extracorporeal membranous oxygenation (ECMO).
  Interventions: Behavioral: Mixed Reality (MR)
- Control (Active Comparator): In the control group, there will be no headset, no heat lamps, and no weighted vest and the participant will rely on their imagination to embody the teenager while lying in the simulation room bed while being consented for the same procedure as the MR group.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Mixed Reality (MR) — Mixed Reality simulation of medical crisis scenarios.
  MR headset - a device that the participants will wear over their head and eyes and will add holographic elements to a live view of workplace training scenario
  Arms: Mixed Reality Group
Behavioral: Control — Tradition simulation of medical crisis scenarios.
  Arms: Control

SUMMARY:
This is a quantifiable study evaluating the ability of a mixed reality (MR), immersive simulation experience to evoke empathy in anesthesiology trainees. Quantitative methodologies will be employed using standardized questionnaires including the The Jefferson Scale of Physician Empathy for Health Professions Students, (HP-version). Trainees will assess their preliminary, baseline empathy using the Jefferson Scale and after the simulation and debrief, will reassess empathy scores, once again using the Jefferson Scale. A satisfaction survey to assess simulated patient embodiment as a valuable exercise and contributor to empathy education curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Trainees or personnel working and/or volunteering at Lucile Packard Children's Hospital Stanford / Stanford Health Care facilities
* 18 years and older

Exclusion Criteria:

* a history of severe motion sickness
* currently have nausea
* have a history of seizures
* are uncomfortable wearing a ~7 pound weighted vest.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported empathy from before and after the simulation | baseline, immediately after the intervention
  Measured with Jefferson Scale of Physician Empathy for physicians and other practicing health professionals (HP-Version). The survey contains 20 item with 7-point scale, 1 indicates strongly disagree and 7 indicates strongly agree (a higher number on the scale indicates more agreement).

SECONDARY OUTCOMES:
Satisfaction of Design Features of the Simulation | immediately after the intervention
  Measured by Simulation Design Scale. The simulation design scale consists of 20 items in total. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. The survey contains 20 item with 5-point scale, 1 indicates strongly disagree and 5 indicates strongly agree (a higher number on the scale indicates more agreement).
  In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. The survey contains 20 item with 5-point scale, 1 indicates not important and 5 indicates very important (a higher number on the scale indicates more important).
  In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.
Evaluation of the CHARM system's usability | immediately after simulation
  Measured by System Usability Scale (SUS). The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Evaluation of the CHARM system's ergonomics | immediately after simulation
  Measured by the ISO Ergonomic scale. The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States